CLINICAL TRIAL: NCT04100083
Title: Spironolactone in the Treatment of Hidradenitis Suppurativa: a Prospective, Open-Label Proof-of-Concept and Dose-Ranging Study
Brief Title: Spironolactone for Hidradenitis Suppurativa
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00083948
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Spironolactone; Canrenoic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Active Comparator): Patients taking 50mg Spironolactone
  Interventions: Drug: Spironolactone 50 MG
- Group 2 (Active Comparator): Patients taking 100mg Spironolactone
  Interventions: Drug: Spironolactone 100mg
- Group 3 (Active Comparator): Patients taking 200mg Spironolactone
  Interventions: Drug: Spironolactone 200 mg

INTERVENTIONS:
Drug: Spironolactone 50 MG — Study visit timeline: initial visit [consent and enrollment followed by baseline exam (0 months), 3 months, 6 months, and follow up at 7 months, with optional treatment extension period for up to one year of total treatment during which patients will follow up every 3 months
  The drug will be taken via oral tablets once daily for a duration of 6 months. Patients will be instructed to continue any current treatment regimen for hidradenitis suppurativa that was initiated at least 4 weeks prior to their enrollment in the study. Patients will be instructed to avoid potassium supplements and foods containing high levels of potassium, including salt substitutes, which could potentially lead to hyperkalemia. They will be instructed to avoid medications listed in the exclusion criteria.
  Arms: Group 1
Drug: Spironolactone 100mg — Study visit timeline: initial visit [consent and enrollment followed by baseline exam (0 months), 3 months, 6 months, and follow up at 7 months, with optional treatment extension period for up to one year of total treatment during which patients will follow up every 3 months
  The drug will be taken via oral tablets once daily for a duration of 6 months. Patients will be instructed to continue any current treatment regimen for hidradenitis suppurativa that was initiated at least 4 weeks prior to their enrollment in the study. Patients will be instructed to avoid potassium supplements and foods containing high levels of potassium, including salt substitutes, which could potentially lead to hyperkalemia. They will be instructed to avoid medications listed in the exclusion criteria.
  Arms: Group 2
Drug: Spironolactone 200 mg — Study visit timeline: initial visit [consent and enrollment followed by baseline exam (0 months), 3 months, 6 months, and follow up at 7 months, with optional treatment extension period for up to one year of total treatment during which patients will follow up every 3 months
  The drug will be taken via oral tablets once daily for a duration of 6 months. Patients will be instructed to continue any current treatment regimen for hidradenitis suppurativa that was initiated at least 4 weeks prior to their enrollment in the study. Patients will be instructed to avoid potassium supplements and foods containing high levels of potassium, including salt substitutes, which could potentially lead to hyperkalemia. They will be instructed to avoid medications listed in the exclusion criteria.
  Arms: Group 3

SUMMARY:
The purpose of this study is to evaluate if the drug spironolactone - which is used to treat acne and male pattern hair growth in women - is effective in treating hidradenitis suppurativa in females and which dose of the drug works the best. Participation in this study will take about 4 clinic visits over approximately 7 months with the option to continue for longer if desired.

ELIGIBILITY:
Individuals will be screened for eligibility by a screening visit conducted by named investigators.

Inclusion Criteria To be eligible for the study: (All answers must be "YES" for subject to be eligible.)

1. Subject must have clinically diagnosed hidradenitis suppurativa, with an inadequate response to other treatment modalities, including but not limited to local or systemic antibiotics, immunosuppressive agents, retinoids, biologic therapies, surgical management.
2. Subject disease severity must be classified as 'mild' or more severe on the HS-PGA Scale at screening exam, because subjects classified as 'clear' or 'minimal' on the scale will be unable to achieve the prespecified treatment response.
3. Subject must be a female.
4. Subject must be 18-70 years of age.
5. Women of child-bearing potential must be on effective contraception. Acceptable methods of contraception include oral contraceptive pills (OCPs), hormonal or copper IUDs, contraceptive implants, contraceptive injections, birth control patches, vaginal rings, condom, sponge, diaphragm with spermicide, or prior surgical sterilization.
6. Subject must provide written informed consent prior to any study-related procedures being performed.
7. Subject must be willing to comply with all clinical study procedures.

Exclusion Criteria The presence of the following excludes subjects from the study: (All answers must be "NO" for subject to be eligible.)

1. Subject has previously received spironolactone or another antiandrogenic treatment for hidradenitis suppurativa.
2. The subject is a pregnant or nursing female.
3. Subject is hyperkalemic, defined by a potassium level of greater than 5.1 mEq/liter.
4. Subjects with Addison's disease.
5. Subjects taking eplerenone or other potassium-sparing diuretics, lithium, cholestyramine, ACE inhibitors/angiotensin II antagonists/aldosterone blockers, or NSAIDS.
6. Subjects receiving potassium supplementation.
7. Subjects with history of renal disease or an eFGR < 30.
8. Subjects with acute or chronic liver failure.
9. Subject has an acute psychiatric condition that impairs ability to give consent or follow study protocols.

   * All races and ethnicities will be considered for inclusion in the study.
   * Males will be excluded from this study due to the high incidence of gynecomastia and sexual dysfunction seen in spironolactone use at higher doses in men. It is not routinely used to treat dermatologic conditions in men due to its poor tolerability.
   * Subjects under the age of 18 will not be considered for inclusion in this study. The disease most often manifests during the second and third decades of life, therefore the disorder is far less prevalent in children and adolescents.2

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with 2 grade improvement in Hidradenitis Suppurativa as assessed by physicians global assessment score | Baseline through one year
  The proportion of patients achieving a clinical response - defined as at least a 2-grade improvement in Hidradenitis Suppurativa Physician's Global Assessment (HS-PGA) score relative to baseline at 6 months. HS-PGA is an anchored 6-stage HS-specific physician global assessment scale that was defined for use in a phase-II clinical trial. It is based on the number and type of nodules, abscesses, and fistulas.

SECONDARY OUTCOMES:
Tolerability of spironolactone as measured by incidence of patient reported and physician observed treatment-related adverse events | Baseline through one year
  Adverse effects will define tolerability as Including, but not limited to hyperkalemia, renal insufficiency, menstrual irregularities (metrorrhagia, amenorrhea, breakthrough bleeding), breast tenderness and enlargement, orthostatic hypotension, and changes in libido] and subject self-assessment using the Dermatology Life Quality Index (DLQI) - a validated 10-item dermatology-specific quality of life instrument
Proportion of patients achieving clinical response at month 3 | Baseline through 3 months
  clinical response - defined as at least a 2-grade improvement in Hidradenitis Suppurativa Physician's Global Assessment (HS-PGA) score relative to baseline at 6 months.
  HS-PGA is an anchored 6-stage HS-specific physician global assessment scale that was defined for use in a phase II clinical trial. It is based on the number and type of nodules, abscesses, and fistulas. Its stages are as follows: Clear-No inflammatory or noninflammatory nodules, Minimal-Only the presence of noninflammatory nodules, Mild-<5 inflammatory nodules without abscesses draining fistulas or 1 abscess or draining fistula without additional inflammatory nodules, Moderate-greater than or equal to 5 inflammatory nodules or 1 abscess or draining fistula and greater than or equal to 1 inflammatory nodule or 2-5 abscesses or draining fistulas and <10 inflammatory nodules, Severe-2-5 abscesses or draining fistulas and greater than or equal to 10 inflammatory nodules, Very Severe--5 abscesses or draining fistulas.
Proportion of patients achieving clinical response at any study visits during the optional treatment extension period of up to 1 year | Baseline through one year
  clinical response - defined as at least a 2-grade improvement in Hidradenitis Suppurativa Physician's Global Assessment (HS-PGA) score relative to baseline at 6 months.
  HS-PGA is an anchored 6-stage HS-specific physician global assessment scale that was defined for use in a phase II clinical trial. It is based on the number and type of nodules, abscesses, and fistulas. Its stages are as follows: Clear-No inflammatory or noninflammatory nodules, Minimal-Only the presence of noninflammatory nodules, Mild-<5 inflammatory nodules without abscesses draining fistulas or 1 abscess or draining fistula without additional inflammatory nodules, Moderate-greater than or equal to 5 inflammatory nodules or 1 abscess or draining fistula and greater than or equal to 1 inflammatory nodule or 2-5 abscesses or draining fistulas and <10 inflammatory nodules, Severe-2-5 abscesses or draining fistulas and greater than or equal to 10 inflammatory nodules, Very Severe--5 abscesses or draining fistulas.
Change in patient-reported disease activity | Baseline through one year
  Change will be define from baseline using a 100 mm VAS ranging from 0 mm (no disease activity) and 100 mm (worst disease activity possible),
Comparison between group treatment effects | Baseline through one year
  This will be defined as the estimate of difference in proportion of treatment responders between three treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Elston, MD, Principal Investigator — Medical University of South Carolina

IPD SHARING:
Plan to Share IPD: No